CLINICAL TRIAL: NCT05674890
Title: Comparison of a Novel Head-Mounted Perimeter Versus the Humphrey Field Analyzer
Brief Title: SmartSystem Virtual Reality Headset Perimeter Versus Humphrey HFA-III Perimeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Pouw, MD (Other)
Responsible Party: Sponsor-Investigator, Andrew Pouw, MD, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202206347
Record Dates: First submitted 2023-01-03; First posted 2023-01-09 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: The described study was a validation study comparing a novel testing device to the current clinical standard. The order of testing was randomized, so the design is that of a crossover study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A: HFA followed by SSVR (Other): Patients will have one or both eyes (dependent on inclusion/exclusion criteria) tested with both the Humphrey HFA-III perimeter and the SmartSystem VR headset on the same clinic visit, spaced roughly 10-15 minutes apart. The sequence in which each patient undertakes the two tests will be randomized. Group A includes participants who tested using the HFA, followed by a 15 minute rest period, then tested with the SSVR.
  Interventions: Diagnostic Test: SmartSystem VR Headset perimeter
- Group B: SSVR followed by HFA (Other): Patients will have one or both eyes (dependent on inclusion/exclusion criteria) tested with both the Humphrey HFA-III perimeter and the SmartSystem VR headset on the same clinic visit, spaced roughly 10-15 minutes apart. The sequence in which each patient undertakes the two tests will be randomized. Group B includes participants who tested using the SSVR, followed by a 15 minute rest period, then tested with the HFA.
  Interventions: Diagnostic Test: SmartSystem VR Headset perimeter

INTERVENTIONS:
Diagnostic Test: SmartSystem VR Headset perimeter — Patients will undergo visual field testing with the head-mounted SmartSystem VR Headset perimeter.

SUMMARY:
The goal of this clinical trial is to compare a new device for testing peripheral vision (the SmartSystem virtual reality headset) to the currently most commonly used standard testing device (the Humphrey HFA-III). The main questions this clinical trials aims to answer are:

1. How comparable in performance, accuracy, and patient comfort the SmartSystem VR headset is to the Humphrey HFA-III, and
2. Surveying patients about the perceived ease of use and patient experience with the SmartSystem VR headset, compared to the Humphrey HFA-III.

Participants will be asked to use the SmartSystem VR headset to take an additional visual field test (which takes between 10 to 15 minutes to do) and to take a brief survey about their experience. This will occur on regularly scheduled clinic visits and done in addition to the standard tests and examinations scheduled for that day.

Researchers will compare the patients' test results and survey responses for both the SmartSystem VR headset and the Humphrey HFA-III to see which has more favorable performance, reliability, duration of testing and user experience.

DETAILED DESCRIPTION:
The purpose of this prospective study is to compare the novel SmartSystem VR Headset (M&S Technologies, Niles, IL) to the Humphrey Field Analyzer (Carl Zeiss Meditec Inc., Dublin, CA). Use of the Humphrey Field Analyzer is part of routine clinical care of glaucoma and would be completed regardless of study participation.

The proposed study will be conducted at the University of Iowa Hospitals and Clinics. We estimate 50 subjects will be recruited to participate in the study. Data collected will not include patient identifiers.

The research will involve prospective collection of visual field tests. Patients with suspected, mild, moderate, or severe glaucoma will be included. Clinical data including age, gender, ethnicity, visual acuity, intraocular pressure, severity of disease, Humphrey HFA-III performance, SmartSystem VR Headset performance, and satisfaction survey will be recorded.

Subjects will undergo regular clinical examination, including measurement of visual acuity, intraocular pressure, slit lamp examination by their physician, and visual field testing as indicated. When it comes time to perform visual field testing, subjects will be randomized to complete either the SmartSystem VR Headset visual field test first followed by the Humphrey Field Analyzer visual field test, or vice versa. Visual field tests will be separated by a rest period of 10 to 15 minutes to minimize testing fatigue.

The SmartSystem VR Headset is fit to subjects' head using an adjustable head strap. Once the headset it fit to the subject, a research assistant will send a test to the headset from a bluetooth-connected electronic device using M&S Technologies' secured application platform. Subjects will follow prompts from the SmartSystem VR Headset to complete their visual field test, responding using a handheld "trigger" device. Testing is expected to take approximately 5-15 minutes, depending on the subjects' severity of visual field loss. Following visual field testing using both the SmartySystem VR Headset and Humphrey Field Analyzer, subjects will complete a 13-question satisfaction survey. The total expected time commitment of this study is a 1 to 2 hour visit.

M&S Technologies is the developer of the SmartSystem VR Headset visual field test. As the developers, M&S Technologies maintains a secure, encrypted, HIPAA-compliant database of SmartSystem VR Headset users. This database includes patient profiles containing unique subject IDs (de-identified), birth year (but not specific date), and visual field testing results. Outside of this testing information, M&S Technologies does not have access to any additional patient information.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-100 years of age with suspected, mild, moderate, or severe glaucoma

Exclusion Criteria:

* Non-English speakers, patients with systemic or ocular disease affecting central vision, best corrected visual acuity less than 20/80, neurocognitive or psychiatric disorders that would confound visual field testing, those with physical inability to perform testing, and astigmatism with absolute values greater than 2.00 diopters

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pouw, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quigley HA. Number of people with glaucoma worldwide. Br J Ophthalmol. 1996 May;80(5):389-93. doi: 10.1136/bjo.80.5.389. PMID 8695555
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] Beck RW, Bergstrom TJ, Lichter PR. A clinical comparison of visual field testing with a new automated perimeter, the Humphrey Field Analyzer, and the Goldmann perimeter. Ophthalmology. 1985 Jan;92(1):77-82. doi: 10.1016/s0161-6420(85)34065-4. PMID 3974997
- [Background] Hollander DA, Volpe NJ, Moster ML, Liu GT, Balcer LJ, Judy KD, Galetta SL. Use of a portable head mounted perimetry system to assess bedside visual fields. Br J Ophthalmol. 2000 Oct;84(10):1185-90. doi: 10.1136/bjo.84.10.1185. PMID 11004108
- [Background] Mees L, Upadhyaya S, Kumar P, Kotawala S, Haran S, Rajasekar S, Friedman DS, Venkatesh R. Validation of a Head-mounted Virtual Reality Visual Field Screening Device. J Glaucoma. 2020 Feb;29(2):86-91. doi: 10.1097/IJG.0000000000001415. PMID 31790067
- [Background] Nakai Y, Bessho K, Shono Y, Taoka K, Nakai Y. Comparison of imo and Humphrey field analyzer perimeters in glaucomatous eyes. Int J Ophthalmol. 2021 Dec 18;14(12):1882-1887. doi: 10.18240/ijo.2021.12.11. eCollection 2021. PMID 34926203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 52 subjects (98 eyes) were recruited at the University of Iowa Hospitals and Clinics Department of Ophthalmology and Visual Sciences Glaucoma Service between January 2023 and June 2023.
Pre-assignment Details: Subjects recruited for the present study completed two visual field tests, one with the Smart System VR headset and one with the Humphrey Field Analyzer III. The order of testing was randomized upon study enrollment using a random number generator.
Units Other Than Participants: 98 eyes were tested overall.
Groups:
- Group A: HFA Followed by SSVR: Patients will have one or both eyes (dependent on inclusion/exclusion criteria) tested with both the Humphrey HFA-III perimeter and the SmartSystem VR headset on the same clinic visit, spaced roughly 10-15 minutes apart. The sequence in which each patient undertakes the two tests will be randomized using a random number generator. Group A includes patients who test using the HFA first, followed by a 15 minute rest period, then test with the SSVR.
  SmartSystem VR Headset perimeter: Patients will undergo visual field testing with the head-mounted SmartSystem VR Headset perimeter.
- Group B: SSVR Followed by HFA: Patients will have one or both eyes (dependent on inclusion/exclusion criteria) tested with both the Humphrey HFA-III perimeter and the SmartSystem VR headset on the same clinic visit, spaced roughly 10-15 minutes apart. The sequence in which each patient undertakes the two tests will be randomized using a random number generator. Group B includes patients who test using the SSVR first, followed by a 15 minute rest period, then test with the HFA.
Period: Overall Study
Arm/Group | Group A: HFA Followed by SSVR | Group B: SSVR Followed by HFA
Started (The present study enrolled patients between December 2022 and June 2023. Subjects' participation was limited to the duration of a single clinic appointment. Subjects were not asked to return for study-related testing or follow-up.) | 40; 40 98 eyes were tested overall. | 58; 58 98 eyes were tested overall.
Completed (The target sample size was reached in June 2023.) | 33; 33 98 eyes were tested overall. (Our target number of eyes tested was 80. We recruited 98 total and analyzed 81 due to exclusion of 17 tests.) | 48; 48 98 eyes were tested overall.
Not Completed | 7; 7 98 eyes were tested overall. | 10; 10 98 eyes were tested overall.
Not completed — 5 eyes were excluded due to poor reliability indices | 2 | 3
Not completed — 4 eyes were excluded due to neurocognitive disease interfering with testing capability. | 2 | 2
Not completed — 8 eyes were excluded due to systemic or ocular disease affecting central vision. | 3 | 5

BASELINE CHARACTERISTICS:
Population: Participants were glaucoma patients seen at the University of Iowa Hospitals and Clinics (Iowa City, IA), an academic medical center.
Units Other Than Participants: Eyes
Groups:
- 2-Arm Crossover Study Design: All patients will be in a single arm: patients will have one or both eyes (dependent on inclusion/exclusion criteria) tested with both the Humphrey HFA-III perimeter and the SmartSystem VR headset on the same clinic visit, spaced roughly 10-15 minutes apart. The sequence in which each patient undertakes the two tests will be randomized.
  SmartSystem VR Headset perimeter: Patients will undergo visual field testing with the head-mounted SmartSystem VR Headset perimeter.
Arm/Group | 2-Arm Crossover Study Design
Number analyzed (Participants) | 52
Number analyzed (Eyes) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.70 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Glaucoma Diagnosis [Number; unit: eyes]
  Normal Tension | 31
  Primary Open Angle | 27
  Pseudoexfoliative | 10
  Mixed-Mechanism | 6
  Steroid-Induced | 3
  Chronic Angle Closure | 2
  Aphakic | 2
Glaucoma Severity [Number; unit: eyes]
  Early | 25
  Moderate | 22
  Severe | 34
Spherical Equivalent [Mean (Standard Deviation); unit: Diopters] — Population: We included 40 right eyes and 41 left eyes in our analysis. The total number of eyes was 81 from 45 subjects (both the right and left eye were excluded in 7/52 subjects).
  Diopters
    Right Eye: number analyzed (Participants) | 40
    Right Eye: number analyzed (Eyes) | 40
    Right Eye | -0.72 (1.98)
    Left Eye: number analyzed (Participants) | 41
    Left Eye: number analyzed (Eyes) | 41
    Left Eye | -0.63 (1.85)
    All Eyes: number analyzed (Participants) | 45
    All Eyes | -0.67 (1.90)
Eye Tested [Number; unit: eyes]
  Right Eye | 40
  Left Eye | 41

OUTCOME MEASURES:

1. Primary Outcome: Visual Field Performance Metric #1 - Mean Deviation
Description: Mean deviation indicates how much, on average, an entire visual field deviates from the age-normal value. It is the center-weighted average of the decibel deviations at each point tested in the visual field test. The measurement is reported in decibels.
Time Frame: This measurement will automatically be reported upon conclusion of each visual field test. Visual field testing is estimated to take 5-15 minutes for each visual field test. All testing will occur on the same day within a 1-2 hour period.
Measure: Mean (Standard Deviation); unit: decibels
Units Other Than Participants: Eyes
Groups:
- Single Arm: All patients will be in a single arm: patients will have one or both eyes (dependent on inclusion/exclusion criteria) tested with both the Humphrey HFA-III perimeter and the SmartSystem VR headset on the same clinic visit, spaced roughly 10-15 minutes apart. The sequence in which each patient undertakes the two tests will be randomized.
  SmartSystem VR Headset perimeter: Patients will undergo visual field testing with the head-mounted SmartSystem VR Headset perimeter.
Arm/Group | Single Arm
Number analyzed (Participants) | 45
Number analyzed (Eyes) | 81
decibels
  SSVR MD | -7.17 (6.36)
  HFA MD | -6.88 (4.51)
Statistical Analysis 1: Comparison: Single Arm; Prior to patient enrollment, a power calculation was conducted to assess the ability of our analyses to reliably detect differences between the HFA and SSVR. With a sample size of 80, assumed effect size of 0.15, standard deviation of 0.25, intraclass correlation coefficient of 0.50, and significance level of 0.05, our analysis reaches a power of 0.87; Test type: Equivalence — Any deviation greater that +/- 0.60 (Effect size/Stdev OR 0.15/0.25=0.60) between device means was considered "non-equivalent"; p = 0.297, t-test, 2 sided; Mean Difference (Net) = -0.29, Standard Deviation 2.49

2. Primary Outcome: Visual Field Performance Metric #2 - Pattern Standard Deviation
Description: Pattern standard deviation reflects irregularities in a visual field, such as those caused by localized defects. This metric shows sensitivity losses after adjusting for generalized depression or elevation in the overall hill of vision (e.g. cataracts). The measurement is reported in decibels.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: decibels
Units Other Than Participants: Eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 45
Number analyzed (Eyes) | 81
decibels
  SSVR PSD | 4.26 (2.37)
  HFA PSD | 6.38 (4.51)
Statistical Analysis 1: Comparison: Single Arm; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -2.11, Standard Deviation 2.81

3. Primary Outcome: Visual Field Performance Metric #3 - Test Duration
Description: This metric indicates how long each visual field test took to complete per eye.
Time Frame: These measurements will be derived during data analysis following study completion. The exact study duration is unclear; however, we aim to recruit enough patients to analyze 80 eyes worth of data. We estimate this will take 3-6 months.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 45
Number analyzed (eyes) | 81
seconds
  SSVR Test Duration | 323.44 (72.27)
  HFA Test Duration | 372.20 (61.44)
Statistical Analysis 1: Comparison: Single Arm; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -48.75, Standard Deviation 56.48

4. Secondary Outcome: Visual Field User Experience Question #1 - "How Would You Rate the Comfort of the [Humphrey Field Analyzer/Smart System Virtual Reality Headset]?"
Description: This question will be rated using a Likert scale. Response options will include "very uncomfortable", "uncomfortable", "neutral", "comfortable", and "very comfortable".
Time Frame: Subjects will respond to an approximately 5-10 minute survey upon completion of both visual field tests. The survey will be administered the same day as visual field testing at the conclusion of the estimated 1-2 hour period.
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 52
participants
  SSVR Very Uncomfortable | 0
  SSVR Uncomfortable | 3
  SSVR Neutral | 7
  SSVR Comfortable | 27
  SSVR Very Comfortable | 15
  HFA Very Uncomfortable | 2
  HFA Uncomfortable | 22
  HFA Neutral | 17
  HFA Comfortable | 7
  HFA Very Comfortable | 4

5. Secondary Outcome: Visual Field User Experience Question #2 - "How Hard or Easy Was it to Understand the Instructions Given to You for How to do the Visual Field Test Using the [Humphrey Field Analyzer/Smart System Virtual Reality Headset]?"
Description: This question will be rated using a Likert scale. Response options will include "very hard", "hard", "neutral", "easy", and "very easy".
Time Frame: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 52
participants
  SSVR Very Hard | 0
  SSVR Hard | 0
  SSVR Neutral | 2
  SSVR Easy | 18
  SSVR Very Easy | 32
  HFA Very Hard | 0
  HFA Hard | 2
  HFA Neutral | 9
  HFA Easy | 19
  HFA Very Easy | 22

6. Secondary Outcome: Visual Field User Experience Question #3 - "How Hard or Easy Was it to Use and/or Perform the Visual Field Test Using the [Humphrey Field Analyzer/Smart System Virtual Reality Headset]?"
Description: as for outcome 5
Time Frame: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 52
participants
  SSVR Very Hard | 0
  SSVR Hard | 0
  SSVR Neutral | 5
  SSVR Easy | 19
  SSVR Very Easy | 28
  HFA Very Hard | 5
  HFA Hard | 19
  HFA Neutral | 15
  HFA Easy | 11
  HFA Very Easy | 2

7. Secondary Outcome: Visual Field User Experience Question #4 - "How Much Anxiety or Concern Did You Have About Your Test Performance While Using the [Humphrey Field Analyzer/Smart System Virtual Reality Headset]?"
Description: This question will be rated using a Likert scale. Response options will include "very anxious/concerned", "anxious/concerned", "neutral", "relaxed", and "very relaxed".
Time Frame: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 52
participants
  SSVR Very Anxious | 0
  SSVR Anxious | 6
  SSVR Neutral | 12
  SSVR Relaxed | 24
  SSVR Very Relaxed | 10
  HFA Very Anxious | 1
  HFA Anxious | 21
  HFA Neutral | 13
  HFA Relaxed | 13
  HFA Very Relaxed | 4

8. Secondary Outcome: Visual Field User Experience Question #5 - "Given Instruction and Training, Would You Feel Comfortable Performing Visual Field Testing by Yourself at Home Using the Smart System Virtual Reality Headset?"
Description: Response options will include "yes", "no", and "maybe".
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 52
Participants
  Yes | 40
  No | 3
  Maybe | 9

9. Secondary Outcome: Visual Field User Experience Question #6 - "If the Smart System Virtual Reality Headset Were Available for Home Use, Would You Use it?"
Description: Response options will include "yes", "no", and "maybe".
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 52
Participants
  Yes | 36
  No | 5
  Maybe | 11

10. Secondary Outcome: Visual Field User Experience Question #7 - "Which Visual Field Test Would You Rather Use at Follow-up Visits?"
Description: Response options will include "Humprey Field Analyzer", "Smart System Virtual Reality Headset", and "unsure".
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 52
Participants
  SSVR | 46
  HFA | 2
  Unsure | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study, from December 2022 to June 2023. Individual participants were monitored for the duration of their clinical appointments, approximately 1-2 hours.
Description: The device tested poses no risk to the subjects tested.
Groups:
- Group A: HFA Followed by SSVR: Patients will have one or both eyes (dependent on inclusion/exclusion criteria) tested with both the Humphrey HFA-III perimeter and the SmartSystem VR headset on the same clinic visit, spaced roughly 10-15 minutes apart. The sequence in which each patient undertakes the two tests will be randomized. Group A includes participants who tested using the HFA first, followed by a 15 minute rest period, then tested with the SSVR.
  SmartSystem VR Headset perimeter: Patients will undergo visual field testing with the head-mounted SmartSystem VR Headset perimeter.
- Group B: SSVR Followed by HFA: Patients will have one or both eyes (dependent on inclusion/exclusion criteria) tested with both the Humphrey HFA-III perimeter and the SmartSystem VR headset on the same clinic visit, spaced roughly 10-15 minutes apart. The sequence in which each patient undertakes the two tests will be randomized. Group B includes participants who tested using the SSVR first, followed by a 15 minute rest period, then tested with the HFA.
  SmartSystem VR Headset perimeter: Patients will undergo visual field testing with the head-mounted SmartSystem VR Headset perimeter.
Arm/Group | Group A: HFA Followed by SSVR | Group B: SSVR Followed by HFA
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/31
Other Adverse Events (participants affected / at risk) | 0/21 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05674890/Prot_SAP_001.pdf